CLINICAL TRIAL: NCT00027781
Title: Open Label Phase II Study of MEN-10755 Administered Every 3 Weeks in Patients With Progressive Hormone Refractory Prostate Cancer
Brief Title: MEN-10755 in Treating Patients With Progressive Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16006-30005; EORTC-16006-30005; MAC-07
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sabarubicin

INTERVENTIONS:
Drug: sabarubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of MEN-10755 in treating patients who have progressive prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the activity of MEN-10755 in patients with progressive hormone-refractory adenocarcinoma of the prostate.
* Determine the rate and duration of objective PSA response in patients treated with this drug.
* Determine the clinical response rate in patients with measurable disease treated with this drug.
* Determine the acute side effects of this drug in these patients.

OUTLINE: This is a multicenter study.

Beginning within 2 weeks after the last PSA measurement, patients receive MEN-10755 IV over 30 minutes on day 1. Treatment repeats every 3 weeks for at least 4 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete or partial response continue to receive additional courses. Patients who achieve stable disease may receive more than 4 courses at the discretion of the investigator.

Patients are followed every 6 weeks until disease progression or initiation of a new therapy.

PROJECTED ACCRUAL: A total of 18-32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hormone-refractory adenocarcinoma of the prostate
* Disease progression while on prior luteinizing hormone-releasing hormone (LHRH) analogues or after orchiectomy and antiandrogens, given concurrently or consecutively
* Disease progression is defined as PSA progression documented by increases in PSA recorded at 2 consecutive measurements over a prior reference value

  * Interval of at least 1 week between the reference value and the first of these two PSA increases
* Continued elevation of PSA for at least 6 weeks after discontinuation of antiandrogens
* Last PSA value at least 5 ng/mL (Hybritech equivalent)
* Must have serum testosterone less than 50 ng/mL and must continue on LHRH agonist therapy if no prior surgical castration
* No symptomatic brain or leptomeningeal metastatic disease

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* ALT/AST no greater than 2.5 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.7 mg/dL
* No uncontrolled hypercalcemia

Cardiovascular:

* No history of severe heart disease
* No myocardial infarction within the past 6 months
* No cardiac insufficiency
* Normal cardiac function by MUGA scan and 12-lead EKG

Other:

* No other prior or concurrent malignancy except basal cell or squamous cell skin cancer
* No uncontrolled systemic nonmalignant disease or infection
* No psychological, familial, or geographical conditions that would preclude compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No prior hormonal therapy except estramustine
* No concurrent estramustine

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy (e.g., for painful bone metastases)

Surgery:

* See Disease Characteristics

Other:

* No other concurrent experimental drugs or investigational therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2001-08; Primary Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Fiedler, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (10):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - CHU de la Timone, Marseille
  - CHU Pitie-Salpetriere, Paris
- Universitaets-Krankenhaus Eppendorf, Hamburg, Germany
- Rabin Medical Center - Beilinson Campus, Petah Tikva, Israel
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Inselspital, Bern, Bern, Switzerland

REFERENCES:
- [Result] Fiedler W, Tchen N, Bloch J, Fargeot P, Sorio R, Vermorken JB, Collette L, Lacombe D, Twelves C; EORTC new drug development group. A study from the EORTC new drug development group: open label phase II study of sabarubicin (MEN-10755) in patients with progressive hormone refractory prostate cancer. Eur J Cancer. 2006 Jan;42(2):200-4. doi: 10.1016/j.ejca.2005.07.030. Epub 2005 Dec 7. PMID 16337787